CLINICAL TRIAL: NCT07373574
Title: Effects of the Dietary Supplements, Congaplex® and Immuplex®, on Age-Related Changes in Fingernail and Hair Health
Brief Title: Effects of Dietary Supplements on Nail and Hair Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Collaborators: UNC Nutrition Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD-01; Pro00088817 (Other: Advarra)
Record Dates: First submitted 2025-09-24; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Nutrient Intake; Nutrient Intake Inadequacy
Keywords: Nutrition; Hair Health; Nail Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Congaplex (Experimental): TP1: 6 capsules/day
  Interventions: Dietary Supplement: Immune Health (Congaplex)
- Immuplex (Experimental): TP2: 6 capsules/day
  Interventions: Dietary Supplement: Immune Health (Immuplex)
- Gastro-Fiber (Active Comparator): AC: 6 capsules/day
  Interventions: Dietary Supplement: Active Control (Gastro-Fiber)

INTERVENTIONS:
Dietary Supplement: Immune Health (Congaplex) — Supplement related to nail, hair, and immune health
  Arms: Congaplex
Dietary Supplement: Active Control (Gastro-Fiber) — Supplement not related to immune, hair, or nail health
  Arms: Gastro-Fiber
Dietary Supplement: Immune Health (Immuplex) — Supplement related to nail, hair, and immune health
  Arms: Immuplex

SUMMARY:
This is a research study conducted by Standard Process, Inc. and the University of North Carolina and Chapel Hill Nutrition Research Institute, which aims to evaluate the effectiveness of nutritional supplementation in improving the health of fingernails and hair. We value your participation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, controlled clinical trial focused on evaluating the effects of two nutritional supplements, Congaplex® (test product 1, TP1) and Immuplex® (TP2), versus an active control (AC) product, Gastro-Fiber®, on the health of fingernails and hair. The study will include a total of 90 participants across 3 arms and use a parallel-group design: 30 participants in TP1 group, 30 participants in TP2 group, and 30 participants in the AC group. The participants and the research personnel will be blind to the treatment. The AC product contains powder in capsules that have an identical size and similar appearance to Congaplex® and Immuplex® supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male adults who are 18 to 75 years of age (inclusive)
2. Display longitudinal (vertical) nail ridges in the absence of other nail abnormalities
3. No cosmetic nail treatments that would mask the natural appearance of the nail plate in the past 6 months (i.e., manicure procedures that smooth the nail surface, nail polish)
4. In good general health (no uncontrolled diseases or conditions) as deemed by the investigator and is able to consume the study product
5. Individuals with childbearing potential must agree to practice an acceptable form of birth control for a certain timeframe prior to the first dose of study product and throughout the study, including:

   1. use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), or hormone implant (e.g., Norplant System), or intrauterine devices (e.g., Mirena); or
   2. use for at least 1 month prior to the first dose of study product: double-barrier method, non-hormonal intrauterine devices (i.e., copper), or complete abstinence from sexual intercourse that may result in pregnancy; or
   3. vasectomy of partner at least 6 months prior to the first dose of study product.

   A participant of childbearing potential must use 1 highly effective contraceptive method during the study or use the double-barrier method during the study. Individuals with the potential to impregnate others must agree to use condoms or other acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that may result in pregnancy is also acceptable.
6. Agree to refrain from treatments listed in Section 8.3 in the defined timeframe.
7. Have maintained stable dietary habits (including supplement intake), exercise habits and lifestyle for the last 3 months prior to screening and agree to maintain dietary and exercise habits and lifestyle throughout the study.
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study as confirmed at the baseline visit (Visit 2)
2. Individuals who have applied cosmetic/topical treatments to fingernails in the past 6 months (i.e., manicures with nail plate filing, nail polish)
3. Individuals who display nail abnormalities indicative of a health condition affecting nail appearance or have been diagnosed with a disease affecting nails (i.e., thickening, discoloration, horizontal nail ridges [Beau's lines])
4. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients
5. Currently has COVID-19 or tests positive for COVID-19 within 28 days prior to baseline visit
6. Individuals opposed to consuming animal products
7. Have a history of uncontrolled hypertension (140/90 or greater mmHg), kidney dysfunction or disease (dialysis or renal failure), hepatic impairment or disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Determine the effects of test products (TP1/2) versus active control (AC) on numbers and severity of longitudinal (vertical) nail ridges | 6 months
  Changes in scores of vertical nail ridge numbers and severity according to Nail Score Chart from baseline to months 3 and 6 of supplementation. Higher number of vertical ridges indicate poorer outcome.
Determine the effects of TP1/2 versus AC on nail biostructure and biochemical composition after 6 months of supplementation | 6 months
  Changes in Raman spectra of fingernail and surround tissue from baseline to month 6 of supplementation

SECONDARY OUTCOMES:
Determine the effects of test products TP1/2 versus AC on density, thickness and pigmentation of hair | 6 months
  Changes in hair density, thickness and pigmentation from baseline to months 3 and 6 of supplementation, measured by trichoscopy. Trichoscopy is a non-invasive procedure that allows examination of the scalp and hair at a high magnification to examine hair and scalp health. This will look at the quality of the hair.
Determine the effects of TP1/2 versus AC on hair biostructure and biochemical compositions after 3 and 6 months of supplementation | 6 months
  Changes in Raman spectra of newly grown parts of nail from baseline to months 3 and 6 of supplementation to compare quality of nail structure
Determine the effects of TP1/2 versus AC on near vision (visual accommodation) | 6 months
  Change in vision and near vision from baseline to months 3 and 6 of supplementation, measured using a Bailey Lovie Chart
Determine the effects of TP1/2 versus AC on the scores of general health questionnaire | 6 months
  Changes in the total scores and subscores of a 36-Item Health Survey Instrument (SF-36) from baseline to months 3 and 6 of supplementation

OTHER OUTCOMES:
Assess the safety and tolerability of TP1/2 and AC in healthy participants | 6 months
  Reports of adverse events
Anthropometrics | 6 months
  Changes in body mass index [BMI] from baseline to 3 months and six months of supplementation
Vitals | 6 months
  Changes in blood pressure [BP] from baseline to 3 and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in blood urea nitrogen (BUN) from baseline to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in triglycerides from baseline to 3 months, and 6 months of supplementation
Hepatic Biomarkers | 6 months
  Changes in alanine aminotransferase (ALT) from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in immunoglobulin E (IgE) from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in total cortisol from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in free triiodothyronine (T3) from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in vitamin D from baseline to 3 months, and 6 months of supplementation.
Cognition Biomarkers | 6 months
  Changes in folate from baseline to 3 months, and 6 months of supplementation.
Polyamine Biomarkers | 6 months
  Changes in spermidine from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-1 from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in autoantibodies against citrullinated and non-citrullinated collagen from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in C-Peptide from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in Creatine Kinase (CK) from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in Creatinine from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in estimated glomerular filtration rate from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in glucose from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in hemoglobin A1C from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in insulin from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in lactate dehydrogenase (LD) from baseline to 3 months, and 6 months of supplementation.
Metabolic Biomarkers | 6 months
  Changes in blood uric acid from baseline to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in total cholesterol from baseline to 3 months, and 6 months of supplementation
Lipid Panel Biomarkers | 6 months
  Changes in low-density lipoprotein (LDL) from baseline to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in high-density lipoprotein cholesterol (HDL-C) from to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in lipoprotein (Lpa) from baseline to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in apolipoprotein (ApoA) from baseline to 3 months, and 6 months of supplementation.
Lipid Panel Biomarkers | 6 months
  Changes in apolipoprotein (ApoB) from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in albumin from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in alkaline phosphatase (ALP) from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in aspartate aminotransferase (AST) from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in C-Reactive protein (CRP) from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in gamma-glutamyl transferase (GGT) from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in total bilirubin from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in globulin from baseline to 3 months, and 6 months of supplementation.
Hepatic Biomarkers | 6 months
  Changes in total protein from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in immunoglobulin M (IgM) from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in immunoglobulin A (IgA) from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in immunoglobulin G (IgG) from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in rheumatoid factor (RF) from baseline to 3 months, and 6 months of supplementation.
Immune Biomarkers | 6 months
  Changes in anti-citrullinated protein antibodies from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in corticosteroid-binding globulin (free cortisol index) from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in dehydroepiandrosterone (DHEA) from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in estradiol from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in sex hormone-binding globulin (SHBG) from baseline to 3 months, and 6 months of supplementation.
Adrenal Hormone Biomarkers | 6 months
  Changes in testosterone from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in free thyroxine (T4) from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in total T3 from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in total T4 from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in thyroid stimulating hormone (TSH) from baseline to 3 months, and 6 months of supplementation.
Thyroid Hormone Biomarkers | 6 months
  Changes in triiodothyronine uptake test from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in ferritin from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in iron from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in chloride from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in phosphorus from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in potassium from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in sodium from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in calcium from baseline to 3 months, and 6 months of supplementation.
Vitamins and Mineral | 6 months
  Changes in magnesium from baseline to 3 months, and 6 months of supplementation.
Cognition Biomarkers | 6 months
  Changes in homocysteine from baseline to 3 months, and 6 months of supplementation.
Cognition Biomarkers | 6 months
  Changes in vitamin B12 from baseline to 3 months, and 6 months of supplementation.
Polyamine Biomarkers | 6 months
  Changes in spermine from baseline to 3 months, and 6 months of supplementation.
Polyamine Biomarkers | 6 months
  Changes in histamine from baseline to 3 months, and 6 months of supplementation.
Polyamine Biomarkers | 6 months
  Changes in putrescine from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-1 receptor antagonist protein (IL-1RN) from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-6 from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-8 from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-13 from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in INF alpha from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IL-18 from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in IFN beta from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in TGF beta from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in TNF from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in serum amyloid A from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in serum tau from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in neurofilament light from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in S100B from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in GFAP from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in NLR from baseline to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in biomarkers from CRP to 3 months, and 6 months of supplementation.
Inflammation Biomarkers | 6 months
  Changes in CAR from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in fibronectin from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in vimentin from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in NSE from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in ICAM from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in actin from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in zonulin from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in MYH7 from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in myoglobin from baseline to 3 months, and 6 months of supplementation.
Other Biomarkers | 6 months
  Changes in troponin from baseline to 3 months, and 6 months of supplementation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozeren E. Is C-reactive protein-albumin ratio or neutrophil-lymphocyte ratio a better indicator to predict in-hospital mortality in traumatic brain injury? Ulus Travma Acil Cerrahi Derg. 2022 Oct;28(10):1482-1487. doi: 10.14744/tjtes.2022.00794. PMID 36169474
- [Background] Baccaglini L, Theriaque DW, Shuster JJ, Serrano G, Lalla RV. Validation of anamnestic diagnostic criteria for recurrent aphthous stomatitis. J Oral Pathol Med. 2013 Apr;42(4):290-4. doi: 10.1111/jop.12015. Epub 2012 Oct 27. PMID 23106421
- [Background] Karincaoglu Y, Batcioglu K, Erdem T, Esrefoglu M, Genc M. The levels of plasma and salivary antioxidants in the patient with recurrent aphthous stomatitis. J Oral Pathol Med. 2005 Jan;34(1):7-12. doi: 10.1111/j.1600-0714.2004.00253.x. PMID 15610400
- [Background] Arikan S, Durusoy C, Akalin N, Haberal A, Seckin D. Oxidant/antioxidant status in recurrent aphthous stomatitis. Oral Dis. 2009 Oct;15(7):512-5. doi: 10.1111/j.1601-0825.2009.01580.x. PMID 19761497
- [Background] Edgar NR, Saleh D, Miller RA. Recurrent Aphthous Stomatitis: A Review. J Clin Aesthet Dermatol. 2017 Mar;10(3):26-36. Epub 2017 Mar 1. PMID 28360966
- [Background] Tappuni AR, Kovacevic T, Shirlaw PJ, Challacombe SJ. Clinical assessment of disease severity in recurrent aphthous stomatitis. J Oral Pathol Med. 2013 Sep;42(8):635-41. doi: 10.1111/jop.12059. Epub 2013 Mar 19. PMID 23509958
- [Background] Sanchez-Bernal J, Conejero C, Conejero R. Recurrent Aphthous Stomatitis. Actas Dermosifiliogr (Engl Ed). 2020 Jul-Aug;111(6):471-480. doi: 10.1016/j.ad.2019.09.004. Epub 2020 May 22. English, Spanish. PMID 32451064
- [Background] Chang H, Johnson E, Khoo C, Wang W, Gu L. Cranberry Juice Polyphenols Inhibited the Formation of Advanced Glycation End Products in Collagens, Inhibited Advanced Glycation End Product-Induced Collagen Crosslinking, and Cleaved the Formed Crosslinks. J Agric Food Chem. 2022 Dec 14;70(49):15560-15569. doi: 10.1021/acs.jafc.2c06502. Epub 2022 Dec 1. PMID 36455288
- [Background] Haus JM, Carrithers JA, Trappe SW, Trappe TA. Collagen, cross-linking, and advanced glycation end products in aging human skeletal muscle. J Appl Physiol (1985). 2007 Dec;103(6):2068-76. doi: 10.1152/japplphysiol.00670.2007. Epub 2007 Sep 27. PMID 17901242
- [Background] Aggarwala KRG. Ocular Accommodation, Intraocular Pressure, Development of Myopia and Glaucoma: Role of Ciliary Muscle, Choroid and Metabolism. Med Hypothesis Discov Innov Ophthalmol. 2020;9(1):66-70. Epub 2020 Jan 5. PMID 31976346
- [Background] Kuzuhara A, Fujiwara N, Hori T. Analysis of internal structure changes in black human hair keratin fibers with aging using Raman spectroscopy. Biopolymers. 2007 Oct 5-15;87(2-3):134-40. doi: 10.1002/bip.20805. PMID 17626296
- [Background] Brito ALB, Bruggen C, Ildiz GO, Fausto R. Investigation of menopause-induced changes on hair by Raman spectroscopy and chemometrics. Spectrochim Acta A Mol Biomol Spectrosc. 2022 Jul 5;275:121175. doi: 10.1016/j.saa.2022.121175. Epub 2022 Mar 21. PMID 35344858
- [Background] Jain N, Doshi B, Khopkar U. Trichoscopy in alopecias: diagnosis simplified. Int J Trichology. 2013 Oct;5(4):170-8. doi: 10.4103/0974-7753.130385. PMID 24778525
- [Background] Park AM, Khan S, Rawnsley J. Hair Biology: Growth and Pigmentation. Facial Plast Surg Clin North Am. 2018 Nov;26(4):415-424. doi: 10.1016/j.fsc.2018.06.003. Epub 2018 Aug 16. PMID 30213423
- [Background] Gniadecka M, Faurskov Nielsen O, Christensen DH, Wulf HC. Structure of water, proteins, and lipids in intact human skin, hair, and nail. J Invest Dermatol. 1998 Apr;110(4):393-8. doi: 10.1046/j.1523-1747.1998.00146.x. PMID 9540981
- [Background] Fawcett RS, Linford S, Stulberg DL. Nail abnormalities: clues to systemic disease. Am Fam Physician. 2004 Mar 15;69(6):1417-24. PMID 15053406
- [Background] Yin J, Ibrahim S, Petersen F, Yu X. Autoimmunomic Signatures of Aging and Age-Related Neurodegenerative Diseases Are Associated With Brain Function and Ribosomal Proteins. Front Aging Neurosci. 2021 May 28;13:679688. doi: 10.3389/fnagi.2021.679688. eCollection 2021. PMID 34122052
- [Background] Hanlon PR, Robbins MG, Scholl C, Barnes DM. Aqueous extracts from dietary supplements influence the production of inflammatory cytokines in immortalized and primary T lymphocytes. BMC Complement Altern Med. 2009 Dec 14;9:51. doi: 10.1186/1472-6882-9-51. PMID 20003431
- [Background] Juszczak E, Altman DG, Hopewell S, Schulz K. Reporting of Multi-Arm Parallel-Group Randomized Trials: Extension of the CONSORT 2010 Statement. JAMA. 2019 Apr 23;321(16):1610-1620. doi: 10.1001/jama.2019.3087. PMID 31012939
- [Background] Blumberg J. Nutritional needs of seniors. J Am Coll Nutr. 1997 Dec;16(6):517-23. PMID 9430078
- [Background] Ramaa CS, Shirode AR, Mundada AS, Kadam VJ. Nutraceuticals--an emerging era in the treatment and prevention of cardiovascular diseases. Curr Pharm Biotechnol. 2006 Feb;7(1):15-23. doi: 10.2174/138920106775789647. PMID 16472130
- [Background] Sachdeva V, Roy A, Bharadvaja N. Current Prospects of Nutraceuticals: A Review. Curr Pharm Biotechnol. 2020;21(10):884-896. doi: 10.2174/1389201021666200130113441. PMID 32000642
- [Background] Bruins MJ, Van Dael P, Eggersdorfer M. The Role of Nutrients in Reducing the Risk for Noncommunicable Diseases during Aging. Nutrients. 2019 Jan 4;11(1):85. doi: 10.3390/nu11010085. PMID 30621135
- [Background] Odden, M. C. et al. The impact of the aging population on coronary heart disease in the United States. Am J Med 124, 827-833 e825 (2011). https://doi.org:10.1016/j.amjmed.2011.04.010
- [Background] Musillo, C. et al. Natural products improve healthspan in aged mice and rats: A systematic review and meta-analysis. Neurosci Biobehav Rev 121, 89-105 (2021). https://doi.org:10.1016/j.neubiorev.2020.12.001